CLINICAL TRIAL: NCT06238999
Title: Clinical Evaluation of a New Flowable Composite for Direct Restorative Treatment of Non-carious Cervical Lesions: A Prospective Randomized Split-mouth Study
Brief Title: Split-mouth Study of a New Flowable Composite in Non-carious Cervical Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTCS 36427036
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-07

CONDITIONS: Non-carious Cervical Lesions

STUDY DESIGN:
Intervention Model Description: Split-Mouth Design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test goup TM Flow (Experimental): The newly developed flowable composite TM Flow will be used for the restoration of NCCLs in the test group. The treatment workflow is very similar to other flowable composites.
  Interventions: Device: Restoration of non-carious cervical lesions
- Control group Tetric EvoFlow (Active Comparator): The well-established Tetric EvoFlow will be used for the restorations of NCCLs in the control group.
  Interventions: Device: Restoration of non-carious cervical lesions

INTERVENTIONS:
Device: Restoration of non-carious cervical lesions — Non-carious cervical lesions will be treated with the experimental TM Flow or the well-established Tetric EvoFlow. The treatment workflow is very similar to other flowable composites.

SUMMARY:
The overall objective of this clinical investigation is to evaluate the clinical safety and performance of the new flowable composite TM Flow for treatment of non-carious cervical lesions. Each participant receives two different fillings (test- and control material) in two different teeth. The fillings are assessed according to selected FDI criteria at baseline (7-10 days after filling placement) and after 1, 6, 12, 24, 36 and 60 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent signed by the subject
* Age: 18-65 years
* 2 NCCL needing treatment, comparable in extend and size, preferably located in different quadrants
* Vital teeth, regular sensitivity
* Sufficient language skills
* No active periodontitis
* Preoperative VAS values < 3 regarding tooth sensitivity on biting. Tooth sensitivity on temperature or touching (tooth brushing, probing) originating in the area of the NCCL is accepted.
* Subject wishes to have a restoration as part of the study (written declaration of consent after detailed explanation)

Exclusion Criteria:

* Not completed hygiene phase or poor oral hygiene
* Sufficient isolation of the cavity not possible
* Patients with a proven allergy to one of the ingredients (methacrylates)
* Patients with severe systemic diseases
* Periodontally insufficient dentition
* Pregnancy
* Part of the development project team of TM Flow
* Staff of the study management team
* Staff of the internal clinic

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-02-20 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2029-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Ivoclar Vivadent AG, Schaan, Liechtenstein, Liechtenstein

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Teeth
Period: Overall Study
Arm/Group | Test goup TM Flow | Control group Tetric EvoFlow
Started | 66; 66 Teeth | 66; 66 Teeth
Completed | 66; 66 Teeth | 66; 66 Teeth
Not Completed | 0; 0 Teeth | 0; 0 Teeth

BASELINE CHARACTERISTICS:
Units Other Than Participants: Teeth
Groups:
- Total: Total of all reporting groups
Arm/Group | Test goup TM Flow | Control group Tetric EvoFlow | Total
Number analyzed (Participants) | 66 | 66 | 198
Number analyzed (Teeth) | 66 | 66 | 132
Age, Customized [Number; unit: Participants]
  number analyzed (Participants) | 66 | 66 | 66
  <= 18 years | 0 | 0 | 0
  18 to 65 years | 66 | 66 | 66
  > 65 years | 0 | 0 | 0
Sex/Gender, Customized [Number; unit: Participants]
  number analyzed (Participants) | 66 | 66 | 66
  Female | 15 | 15 | 15
  Male | 51 | 51 | 51
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Hypersensitivity
Description: assessed by tests with thermal stimuli and occlusal forces (during biting) determined by VAS (Visual Analog Scale, 0 "No pain at all" - 10 "The worst pain imaginable") following the FDI criteria on a scale from 1 "very good" to 5 "unacceptable" FDI 1: no complaint FDI 2: minor complaint FDI 3: distinct pain FDI 4: persistent pain for prolonged period of time FDI 5: treatment unavoidable
Time Frame: 1 month
Measure: Number; unit: Teeth
Units Other Than Participants: Teeth
Arm/Group | Test goup TM Flow | Control group Tetric EvoFlow
Number analyzed (Participants) | 66 | 66
Number analyzed (Teeth) | 66 | 66
Teeth
  FDI Score 1 | 66 | 66
  FDI Score 2-5 | 0 | 0

2. Secondary Outcome: Evaluation of Functional (e.g. Fracture of the Material and Retention), Biological (e.g. Caries at Restoration Margins) and Aesthetic (e.g. Color Match) Properties of the Restorations
Description: will be assessed acooriding to FDI criteria
Time Frame: 5 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 Month Recall
Arm/Group | Test goup TM Flow | Control group Tetric EvoFlow
All-Cause Mortality (participants affected / at risk) | 0/66 | 0/66
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/66
Other Adverse Events (participants affected / at risk) | 0/66 | 0/66

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/99/NCT06238999/Prot_SAP_002.pdf